CLINICAL TRIAL: NCT00002805
Title: Acute Myeloid Leukemia Salvage Therapy for Patients in First Relapse or Who Fail to Achieve an Initial Remission or Who Develop AML as a Second Malignant Neoplasm
Brief Title: Combination Chemotherapy in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2951; CCG-2951; CDR0000064907 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cladribine; Cytarabine; Etoposide; Methotrexate; Mitoxantrone; Hydrocortisone; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Induction will consist of one course of cytarabine and mitoxantrone. Patients achieving a complete or partial response by the end of induction will start intensification. Intensification will consist of one course of chemotherapy (Cytarabine (Ara-C), Etoposide (VP-16), Filgrastim (G-CSF)). Patients who do not attain a CNS remission following the completion of intensification therapy, or who develop recurrence of CNS disease and have not previously received radiation therapy involving the central nervous system should receive craniospinal radiotherapy. Continuation Therapy: cladribine (2CdA), Etoposide.
  Interventions: Biological: filgrastim; Drug: cladribine; Drug: cytarabine; Drug: etoposide; Drug: methotrexate; Drug: mitoxantrone hydrochloride; Drug: therapeutic hydrocortisone; Procedure: allogeneic bone marrow transplantation; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF; Neupogen; NSC-614629
Drug: cladribine
  Other Names: Leustatin; 2CdA; 2-Chlorodeoxyadenosine
Drug: cytarabine
  Other Names: Ara-C; Cytosine Arabinoside; Cytosar-U
Drug: etoposide
  Other Names: VP-16; VePesid; NSC-141540
Drug: methotrexate
  Other Names: MTX; NSC-740
Drug: mitoxantrone hydrochloride
  Other Names: Novantrone; NSC-301739
Drug: therapeutic hydrocortisone
  Other Names: Hydrocortisone Sodium Succinate; NSC-10483
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients with acute myeloid leukemia or myelodysplastic syndrome in first relapse or who did not achieve first remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity, remission rate, event-free survival, and overall survival following induction with cytarabine/mitoxantrone (ARA-C/DHAD), intensification with ARA-C and etoposide (VP-16), and consolidation with cladribine (2-CdA) and VP-16 in patients with acute myeloid leukemia (AML) that is secondary, in first relapse, or has failed initial remission induction therapy. II. Compare the remission induction rate and event-free survival on this trial with prior second-line studies (i.e., protocols CCG-243, CCG-201, and CCG-261P). III. Compare survival of patients on this trial with the survival of patients relapsing or failing to achieve an initial complete remission (CR) on previous front-line AML trials (i.e., protocols CCG-251, CCG-213, CCG-2861, and CCG-2891). IV. Determine the frequency and prognostic significance of mdr1 gene expression and p53, topoisomerase II, and deoxycytidine kinase gene mutations in these patients. V. Determine the disease-free and overall survival of patients achieving a CR on this study in relation to the post-intensification therapy received (i.e., bone marrow transplantation, chemotherapy, or no further therapy). VI. Determine the frequency and degree of abnormal cardiac function on echocardiogram or MUGA at 1 and 5 years in patients treated with mitoxantrone following anthracycline therapy during initial treatment. VII. Provide a control arm evaluating the safety of using phase I or II agents in an "upfront window" approach planned for future CCG studies. VIII. Determine the toxicity, remission rate, event-free survival, and overall survival in patients who fail to achieve a CR with ARA-C/DHAD induction and are then treated with 2-CdA/VP-16. IX. Determine the biologic characteristics, toxicity, remission rate, event-free survival, and overall survival following this treatment regimen in patients who develop AML as a second malignancy.

OUTLINE: Patients who do not achieve M1/M2a marrow following Induction proceed to Salvage Induction; all others proceed to Intensification. Patients receive Consolidation therapy on Regimen A, B, or C according to the investigator's choice. The following acronyms are used: ARA-C Cytarabine, NSC-63878 2-CdA Cladribine (2-Chlorodeoxyadenosine), NSC-105014 DHAD Mitoxantrone, NSC-301739 G-CSF Filgrastim, NSC-614629 HC Hydrocortisone, NSC-10483 HD High Dose MTX Methotrexate, NSC-740 PBSC Peripheral Blood Stem Cells TBI Total-Body Irradiation TIT Triple Intrathecal Therapy (IT ARA-C/IT HC/IT MTX) VP-16 Etoposide, NSC-141540 INDUCTION: 2-Drug Combination Chemotherapy plus CNS Prophylaxis/Therapy. ARA-C/DHAD; G-CSF; plus IT ARA-C and, if CNS disease at entry, TIT. SALVAGE INDUCTION: 2-Drug Combination Chemotherapy. 2-CdA/VP-16. INTENSIFICATION: 2-Drug Combination Chemotherapy followed, as indicated, by Radiotherapy. HD ARA-C/VP-16; followed, in patients with persistent CNS disease, CNS relapse, or chloromas, by irradiation using megavoltage equipment (minimum Co60 and maximum 6 MV x-rays or electrons). CONSOLIDATION: Regimen A: 2-Drug Combination Chemotherapy. 2-CdA/VP-16. Regimen B: Myeloablative Chemoradiotherapy followed by Hematopoietic Rescue. TBI (equipment unspecified) with electron boosts to the testes, chest, extramedullary sites, and, if indicated, craniospinal region; VP-16; followed by allogeneic or autologous bone marrow or PBSC. Regimen C: No further therapy.

PROJECTED ACCRUAL: A total of 90 patients will be entered. The study may be closed if there are 7 or more deaths in the first 45 patients who complete Intensification.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myeloid leukemia (AML) or myelodysplastic syndrome in one of the following categories: In first relapse Failed to achieve initial complete remission Newly diagnosed secondary AML eligible Required bone marrow status: Greater than 25% blasts (M3) OR Persistent abnormal clone on cytogenetics and 5-25% blasts (M2) No Fanconi's anemia

PATIENT CHARACTERISTICS: Age: Under 22 Performance status: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 times normal AST or ALT less than 4.0 times normal Renal: Creatinine no greater than 1.5 times normal OR Creatinine clearance or GFR greater than 70 mL/min per 1.73 square meters or GFR in equivalent institutional normal range Cardiovascular: Shortening fraction greater than 27% by echocardiogram or in institutional normal range OR Ejection fraction greater than 47% by radionuclide angiogram

PRIOR CONCURRENT THERAPY: No more than 1 prior treatment No prior salvage therapy No prior mitoxantrone

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 1997-08; Primary Completion 2001-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Estimate second remission rate and survival rate | 3 years

SECONDARY OUTCOMES:
Evaluate the mortality of the start of VP-16/Ara-C intensification | 45 days
Compare outcomes by the ethnicity and gender
  Compare outcomes by the ethnicity (and gender) in study CCG-2951, and will control for ethnicity in multivariate models comparing the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Wells, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (38):
- United States (35):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia